CLINICAL TRIAL: NCT03448458
Title: Molecular Imaging With Ga-68 DOTATATE PET to Investigate Neuroendocrine Differentiation in Prostate Cancer Patients
Brief Title: Gallium Ga 68-DOTATATE PET/CT in Diagnosing Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mehmet Bilen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00099167; NCI-2017-02055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4165-17 (Other: Winship Cancer Institute)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ga(III)-DOTATOC; gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gallium Ga 68-DOTATATE PET/CT (Experimental): Patients receive gallium Ga 68-DOTATATE IV. Within 55-70 minutes, patients undergo PET (positron emission tomography)/CT (computed tomography).
  Interventions: Procedure: CT (Computed Tomography); Drug: Gallium Ga 68-DOTATATE; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: CT (Computed Tomography) — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT scan
Drug: Gallium Ga 68-DOTATATE — Given IV
  Other Names: 68Ga-DOTATATE; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies how well gallium Ga 68-DOTATATE positron emission tomography (PET)/computed tomography (CT) works in treating patients with castration resistant prostate cancer that has spread to other placed in the body. Gallium Ga 68-DOTATATE PET/CT may help doctors to identify those patients with early neuroendocrine transdifferentiation and who are at greater risk for poor outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Establish the feasibility of using gallium Ga 68-DOTATATE (68Ga-DOTATATE) PET as a predictive imaging biomarker for neuroendocrine transdifferentiation in prostate cancer.

SECONDARY OBJECTIVE:

Correlate progression of disease with degree of uptake on 68Ga-DOTATATE PET examination.

OUTLINE:

Patients receive gallium Ga 68-DOTATATE intravenously (IV). Within 55-70 minutes, patients undergo PET/CT.

After completion of study, patients are followed up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic castration resistant prostate carcinoma with skeletal, visceral and/or nodal involvement
* Ability to lie still for PET scanning
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients less than 18 years of age
* Patients without metastatic castration resistant prostate carcinoma with skeletal, visceral and/or nodal involvement
* Inability to lie still for PET scanning
* Patients unable to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Asim Bilen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gallium Ga 68-DOTATATE PET/CT
Started | 17
Completed | 16
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gallium Ga 68-DOTATATE PET/CT
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Gallium Ga 68-DOTATATE Uptake
Description: The number of participants with uptake in each type of lesion will be reported. Will be summarized using descriptive statistics. The inter-rater agreement will be assessed by Kappa statistics or intra-class correlation coefficient. The degree of uptake will be plotted against length of time to progress, and the association will be described by Spearman correlation coefficient with 95% confidence interval (CI). In addition, will dichotomize degree of update by median and defined it as high vs. low, and apply Wilcoxon rank sum test or Fisher exact test wherever appropriate.
Time Frame: During PET/CT scan, up to 2 hours
Population: One patient was subsequently found to have an additional metastatic pulmonary squamous cell carcinoma and was excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gallium Ga 68-DOTATATE PET/CT
Number analyzed (Participants) | 16
Participants
  Bone and visceral/nodal lesions | 11
  Only bone lesions | 4
  Only nodal disease | 1

2. Secondary Outcome: Progression Free Survival
Description: Will be associated with 68Ga-DOTATATE uptake. Will be described by Kaplan-Meier method along log-rank p-value.
Time Frame: Date of enrollment to date of progression (radiographic progression or clinical deterioration) or death, or last follow up if event free, assessed up to 36 months
Population: In total, 17 patients were recruited and received at least one [68Ga]Ga-DOTATATE PET-CT. One patient was subsequently found to have an additional metastatic pulmonary squamous cell carcinoma and was excluded from this analysis
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Gallium Ga 68-DOTATATE PET/CT
Number analyzed (Participants) | 16
months
  Marked Ga-DOTATATE uptake found in 7 of 16 patients analyzed and with a Gleason score range of 7-9: number analyzed (Participants) | 6
  Marked Ga-DOTATATE uptake found in 7 of 16 patients analyzed and with a Gleason score range of 7-9 | 8.1 [1.7 to 21.3]
  Moderate Ga-DOTATATE uptake with a Gleason score of 9: number analyzed (Participants) | 7
  Moderate Ga-DOTATATE uptake with a Gleason score of 9 | 13.3 [2.9 to 20.6]
  Mild Ga-DOTATATE uptake with a Gleason score range of 7-8: number analyzed (Participants) | 3
  Mild Ga-DOTATATE uptake with a Gleason score range of 7-8 | 36 [36 to 36]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Gallium Ga 68-DOTATATE PET/CT
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03448458/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03448458/ICF_000.pdf